CLINICAL TRIAL: NCT00028353
Title: A Chemoprevention Study of an Investigational Drug in Men With High Grade Prostate Intraepithelial Neoplasia (PIN)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GTx (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 211
Record Dates: First submitted 2001-12-22; First posted 2001-12-24 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Prostatic Intraepithelial Neoplasia
Keywords: PIN; High Grade Prostate Intraepithelial Neoplasia (PIN)
MeSH Terms: conditions — Prostatic Intraepithelial Neoplasia | interventions — Toremifene

INTERVENTIONS:
Drug: GTX-006 (Acapodene)

SUMMARY:
If you are a male 30 years of age or older and have a positive diagnosis of high grade (II or III) prostate Intraepithelial Neoplasia (PIN) or have had an abnormal/suspicious prostate biopsy, you may be eligible for this study. This is a study of an investigational medication that may reduce high grade PIN and prevent the occurrence of prostate cancer. This study is currently enrolling up to 500 men at approximately 60 locations in the United States.

DETAILED DESCRIPTION:
High grade PIN is the development of precancerous, abnormal tissue of the prostate gland that puts men at high risk of developing prostate cancer. This study will take one year of participation with clinic visits every three months. There will be two prostate biopsies during the study, at six and twelve months. If qualified to participate, you will be randomly assigned to one of four treatment groups. Three out of four groups are varying doses of the study medication and the other is the placebo group (like a sugar pill).

ELIGIBILITY:
* Must have confirmed high grade PIN on prostate biopsy within past 6 months.
* Must have a serum PSA <12 ng/ml.
* Can not have prostate cancer.
* Have significant ocular opacities.
* Can not take finasteride or other testosterone like supplement.

Min Age: 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2001-04; Study Completion 2003-07

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - Private Practice, Huntsville, Alabama
  - Arkansas Urology Associates, Little Rock, Arkansas
  - South Florida Medical Research, Aventura, Florida
  - UroSearch, Leesburg, Florida
  - The Urology Center of Florida Inc., Ocala, Florida
  - UroSearch, Ocala, Florida
  - Dr. Byron Hodge, Orlando, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Sandy Springs Urology, P.C., Atlanta, Georgia
  - North Idaho Urology, Couer D'Alene, Idaho
  - Wishard Memorial Hospital, Indianapolis, Indiana
  - Mid Atlantic Clinical Research, Rockville, Maryland
  - Newton Wellesley Urology, Newton, Massachusetts
  - Private Practice, Las Vegas, Nevada
  - Medical & Clinical Research Associates, Bay Shore, New York
  - Clinical Research of Westchester, New Rochelle, New York
  - Columbia University, New York, New York
  - Private Practice, Staten Island, New York
  - Salem Research Group, Inc., Winston-Salem, North Carolina
  - Tri-State Urologic Services, Cincinnati, Ohio
  - Urologic Surgery, P.C, Bala-Cynwyd, Pennsylvania
  - Urology Associates of Lancaster, Lancaster, Pennsylvania
  - Urology San Antonio Research, San Antonio, Texas
  - Seattle Urological Associates, Seattle, Washington
  - Madigan Army Medical Center, Tacoma, Washington

REFERENCES:
- See also: Related Info — http://www.gtxinc.com